CLINICAL TRIAL: NCT01304784
Title: A Phase 1 and Pharmacologic Study of MM-111 in Combination With Multiple Treatment Regimens in Patients With Advanced HER2 Positive Solid Tumors
Brief Title: A Study of MM-111 in Combination With Multiple Treatments in Patients With HER2 Positive Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-111-01-01-03
Record Dates: First submitted 2011-02-17; First posted 2011-02-25 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: HER-2 Gene Amplification
Keywords: Solid tumors; Failed at least one line of standard therapy
MeSH Terms: interventions — Cisplatin; Capecitabine; Trastuzumab; MM-111; Lapatinib; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental): Regimen follows a 3-week treatment cycle.
  Cisplatin 80mg/m2 given on day 1 by IV infusion over two hours every three weeks.
  Capecitabine 1000 mg/m2 given orally twice daily for fourteen days each 3-week cycle.
  Up to six 3-week cycles of Cisplatin and Capecitabine to be administered. Trastuzumab given as 8 mg/kg loading dose at week 1 over 90 minutes followed by 6 mg/kg every 3 weeks over 30-90 minutes.
  MM-111 will be administered over 90 minutes for the first infusion and then weekly over 60 minutes thereafter.
  Trastuzumab (every 3 weeks) and MM-111 (weekly) will continue until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Cisplatin, Capecitabine, Trastuzumab and MM-111
- Arm 2 (Experimental): Regiment follows a 4-week treatment cycle.
  The following Lapatinib and Trastuzumab regimen will be given in combination with MM-111 in the following order:
  * Trastuzumab 4 mg/kg loading dose week 1 over 90 minutes
  * Followed by Trastuzumab 2 mg/kg weekly thereafter
  * Lapatinib 1000 mg by mouth (PO) daily
  * MM-111 will be administered over 90 minutes for the first infusion and then weekly over 60 minutes thereafter
  Treatment with this regimen will be continued until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Lapatinib +/- Trastuzumab and MM-111
- Arm 3 (Experimental): Regimen follows a 4-week treatment cycle Paclitaxel dosing should begin first dose on cycle 1 day 1. Paclitaxel will be administered at 80 mg/m2 weekly, as an IV infusion over 60 minutes. The infusion should be prepared as directed in the Paclitaxel package insert. All patients receiving Paclitaxel should be premedicated as per the local institutional guidelines.
  Trastuzumab will be administered via IV over 90 minutes at a 4 mg/kg loading dose for the first infusion followed by weekly infusion of 2 mg/kg over 60 minutes thereafter.
  MM-111 will be administered over 90 minutes for the first infusion and then weekly over 60 minutes thereafter.
  Treatment with this regimen will be continued until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Paclitaxel, Trastuzumab and MM-111
- Arm 4 (Experimental): 4-week treatment cycle. Lapatinib given orally. Paclitaxel dosing on cycle 1 day 1. Paclitaxel given at 80 mg/m2 weekly, as an IV infusion over 60 minutes. The infusion should be prepared as directed in the Paclitaxel package insert. All patients receiving Paclitaxel should be premedicated as per the local institutional guidelines.
  Trastuzumab given via IV over 90 minutes at a 4 mg/kg loading dose for the first infusion followed by weekly infusion of 2 mg/kg over 60 minutes thereafter.
  MM-111 given over 90 minutes for the first infusion and then weekly over 60 minutes thereafter.
  Treatment with this regimen will be continued until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Lapatinib, trastuzumab, paclitaxel, and MM-111
- Arm 5 (Experimental): Docetaxel, trastuzumab and MM-111 3-week treatment cycles with therapies given in the following order: 1) docetaxel, 2) trastuzumab, and 3) MM-111
  Docetaxel given as an IV infusion over 60 minutes every three weeks. The infusion should be prepared as directed in the Docetaxel package insert and any institutional guidelines. All patients receiving Docetaxel should be pre-medicated as per the local institutional guidelines.
  The first dose of trastuzumab is a loading dose of 8 mg/kg administered over 90 minutes followed by every three week dosing at 6 mg/kg over 60 minutes via IV infusion.
  The first dose of MM-111 given over 90 minutes followed by 3 week dosing over 60 minutes in the absence of infusion-related reactions
  Interventions: Drug: Docetaxel, trastuzumab and MM-111

INTERVENTIONS:
Drug: Cisplatin, Capecitabine, Trastuzumab and MM-111 — Conventional chemotherapy
  Other Names: Capecitabine = Xeloda; Trastuzumab = Herceptin
  Arms: Arm 1
Drug: Lapatinib +/- Trastuzumab and MM-111 — Conventional chemotherapy
  Other Names: Trastuzumab = Herceptin; Lapatinib = Tykerb
  Arms: Arm 2
Drug: Paclitaxel, Trastuzumab and MM-111 — Conventional chemotherapy
  Other Names: Trastuzumab = Herceptin; Paclitaxel = Taxol
  Arms: Arm 3
Drug: Lapatinib, trastuzumab, paclitaxel, and MM-111 — Conventional chemo
  Other Names: Trastuzumab = Herceptin; Paclitaxel = Taxol; Lapatinib = Tykerb
  Arms: Arm 4
Drug: Docetaxel, trastuzumab and MM-111 — Conventional chemotherapy
  Other Names: Trastuzumab = Herceptin; Docetaxel = Taxotere
  Arms: Arm 5

SUMMARY:
This study is an open-label, dose-escalation study of MM-111 with five different combination treatments with the main goal of determining the safety of MM-111 with each combination.

DETAILED DESCRIPTION:
To determine the MTD and any DLT of MM 111 when administered in combination with either 1) cisplatin, capecitabine, and trastuzumab; 2) lapatinib +/- trastuzumab; 3) paclitaxel and trastuzumab 4) lapatinib, paclitaxel and trastuzumab or 5) docetaxel and trastuzumab in patients with human epidermal growth factor receptor (HER2+) solid tumors

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed advanced cancer that is positive for HER2, either:

  * At least 3+ positive by immunohistochemistry, or
  * Gene amplified positive by fluorescence in situ hybridization (FISH). Chromogenic in situ hybridization (CISH) is acceptable to confirm HER2 positivity if FISH results are not available.
* The patient's cancer must have recurred or progressed following standard therapy or have not responded to standard therapy. (Patients with previously untreated HER2+ metastatic gastric or gastro-esophageal junction cancer can be enrolled onto the cisplatin, capecitabine, and trastuzumab + MM-111 arm of the study.)
* Patients must be ≥ 18 years of age.
* Patients or their legal representatives must be able to understand and sign an informed consent.
* Patients should have evaluable or measurable disease ≥ 1 cm.
* Patients must have ECOG PS ≤ 1 or Karnofsky performance score of ≥ 70.
* Patients must have adequate hematologic status as evidenced by:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelet count ≥ 100,000 platelets/mm3
  * Hemoglobin ≥ 9 g/dL
* For arms 1, 2, 3 and 4 patients must have adequate hepatic function as evidenced by:

  * Serum total bilirubin ≤ 1.5 × the upper limit of normal (ULN)
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 x ULN (5 × ULN is acceptable if liver metastases are present)
* For arm 5 (Docetaxel) patients must have adequate hepatic function as evidenced by:

  * Serum bilirubin within normal limits,
  * AST and/or ALT < 1.5 X ULN and alkaline phosphatase < 2.5 X ULN if concomitantly elevated
* Patients must have adequate renal function as evidenced by:

  * Serum creatinine ≤ 1.5 × ULN
  * Calculated clearance 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Patients must be recovered from the effects of any prior surgery, radiotherapy or other antineoplastic therapy. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v.4.0) up to Grade 1 is acceptable for patients with pre-existing peripheral neuropathy.
* Patients must have a life expectancy of at least 3 months. Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use an effective form of contraception during the study and for 60 days following the last dose of MM-111.

Exclusion Criteria:

* Patients for whom potentially curative antineoplastic therapy is available
* Patients who are pregnant or lactating
* Patients with an active infection or with an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing. (At the discretion of the Investigator, patients with tumor fever may be enrolled.)
* Patients with untreated and/or symptomatic primary or metastatic central nervous system (CNS) malignancies (Patients with CNS metastases who have undergone surgery or radiotherapy, whose disease is stable, and who have been on a stable dose of corticosteroids for at least 2 weeks prior to the first scheduled day of dosing will be eligible for the trial.)
* Patients with known hypersensitivity to any of the components of MM-111 or who have had hypersensitivity reactions to fully human monoclonal antibodies.
* Patients with a known history of hypersensitivity to any of the drug components of a particular regimen.
* Patients who have received other recent antitumor therapy including:
* Investigational therapy administered within the 28 days prior to the first scheduled day of dosing MM-111. Dosing in < 28 days since receiving investigational therapy is acceptable once a time interval equal to at least five half-lives of the investigational agent have passed.
* Any standard chemotherapy or radiation within 14 days (and having passed the time of any actual or anticipated toxicities) prior to the first scheduled dose of MM-111.

There is no necessary washout for trastuzumab. Patients enrolled to the lapatinib-containing arms of the study do not need to have a washout period for lapatinib.

* Patients with New York Heart Association (NYHA) Class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50%
* History of myocardial infarction within 12 months of enrollment
* Uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg)
* Known angina pectoris requiring medication
* Known clinically significant valvular heart disease
* Known history of high-risk arrhythmias
* Known history of congestive heart failure
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Active gastrointestinal bleedingPatients who have received prior maximum cumulative anthracycline doses:

  * doxorubicin or liposomal doxorubicin doses > 360 mg/m2
  * mitoxantrone > 120 mg/m2 and idarubicin > 90 mg/m2
  * epirubicin doses higher than 720 mg/m2
  * Other (e.g., liposomal doxorubicin or other anthracycline equivalent of 360 mg/m2 of doxorubicin)
  * If more than 1 anthracycline has been used, the cumulative dose must not exceed the equivalent of 360mg/m2 of doxorubicin
* Patients with a history of allogeneic transplant. (Patients with a history of autologous bone marrow or stem cell transplant may be enrolled.)
* Patients with known human immunodeficiency virus (HIV), hepatitis B or C. (If patients have previously been treated for hepatitis C and have undetectable viral loads, they can be considered eligible for the trial.)
* Patients with any other medical or psychological condition, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Determine patient's safety (# of adverse events/serious adverse events) and tolerability of MM-111 in combination with multiple treatment regimens | 30 months
  To determine the maximum tolerated dose (MTD) and any dose limiting toxicity (DLT) of MM-111 when administered in combination with either 1. cisplatin, capecitabine, and trastuzumab; 2. lapatinib +/- trastuzumab; 3. paclitaxel and trastuzumab 4. lapatinib, paclitaxel, trastuzumab; or 5. docetaxel and trastuzumab in patients with HER 2 positive solid tumors

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) profile of MM-111 when administered in combination with multiple treatment regimens. The PK profile will help to determine the phase 2 dose | 33 months
  Treatment regimens include either: 1. cisplatin, capecitabine, and trastuzumab; 2. lapatinib +/- trastuzumab; 3. paclitaxel and trastuzumab; 4. lapatinib, paclitaxel, trastuzumab; or 5. docetaxel and trastuzumab in patients with HER2+ solid tumors.
To establish the recommended Phase 2 dose(s) of MM-111 when administered in each of the combinations assessed (based on PK profile, safety data and overall patient tolerability) | 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Richards, MD, Principal Investigator — Tyler Cancer Center
Locations (15):
- United States (15):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology/Hematology, Albany, New York
  - Innovation Center - Kettering Medical Center Health Network, Kettering, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - GHS Institute of Transitional Oncology Research, Greenville, South Carolina
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology PA North/Sammans Cancer Center, Dallas, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Evergreen Hematology and Oncology, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver Cancer Center, Vancouver, Washington